CLINICAL TRIAL: NCT06918275
Title: Efficacy and Safety of V-LocTM 180 Barbed Sutures Compared to Polyglactin 910 Vicryl in Laparoscopic Isthmocele Repair: A Prospective Randomized Study
Brief Title: Laparoscopic Isthmocele Repair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozan Karadeniz, MD, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSCHospital
Record Dates: First submitted 2025-03-28; First posted 2025-04-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Isthmocele
Keywords: isthmocele; laparoscopy; postmenstrual bleeding; V-LocTM 180; Polyglactin 910

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laparoscopic isthmocele repair using V-LocTM 180 barbed suture (Active Comparator): The isthmocele area will be sutured using V-LocTM 180 barbed suture in a continuous, non-locked fashion. The repair was performed using a two-layer closure technique, ensuring precise reapproximation of the myometrial edges without breaching the uterine cavity, followed by closure of the serosal edges.
  Interventions: Procedure: Laparoscopic isthmocele repair using V-LocTM 180 barbed suture
- laparoscopic isthmocele repair using Polyglactin 910 Vicryl sutures (Active Comparator): The isthmocele area will be sutured using Polyglactin 910 Vicryl sutures in a continuous, non-locked fashion. The repair was performed using a two-layer closure technique, ensuring precise reapproximation of the myometrial edges without breaching the uterine cavity, followed by closure of the serosal edges.
  Interventions: Other: Laparoscopic isthmocele repair using Polyglactin 910 vicryl suture

INTERVENTIONS:
Procedure: Laparoscopic isthmocele repair using V-LocTM 180 barbed suture — The standardized surgical steps for the laparoscopic isthmocele repair were as follows; 1) A 30-degree telescope was introduced through a 10 mm trocar at the umbilicus following the establishment of pneumoperitoneum. 2) Three 5 mm trocars were inserted: two in the bilateral lower quadrants and one in the suprapubic region. 3) The bladder was distended with 300 cc of saline infusion to facilitate dissection of the vesicovaginal space and to allow inferior mobilization of the bladder, thereby ensuring optimal visualization of the isthmocele region. Dissection was performed laterally up to the level of the uterine arteries, thereby minimizing the risk of vascular injury. 4) The light source of the laparoscope was deactivated, enabling the identification of the isthmocele region by utilizing the illumination provided by the hysteroscope. 5) Excision of the abnormal tissue was carried out using an ultrasonic energy device (HARMONIC®), guided by the manipulator shaft as a landmark.
  Arms: laparoscopic isthmocele repair using V-LocTM 180 barbed suture
Other: Laparoscopic isthmocele repair using Polyglactin 910 vicryl suture — The standardized surgical steps for the laparoscopic isthmocele repair were as follows; 1) A 30-degree telescope was introduced through a 10 mm trocar at the umbilicus following the establishment of pneumoperitoneum. 2) Three 5 mm trocars were inserted: two in the bilateral lower quadrants and one in the suprapubic region. 3) The bladder was distended with 300 cc of saline infusion to facilitate dissection of the vesicovaginal space and to allow inferior mobilization of the bladder, thereby ensuring optimal visualization of the isthmocele region. Dissection was performed laterally up to the level of the uterine arteries, thereby minimizing the risk of vascular injury. 4) The light source of the laparoscope was deactivated, enabling the identification of the isthmocele region by utilizing the illumination provided by the hysteroscope. 5) Excision of the abnormal tissue was carried out using an ultrasonic energy device (HARMONIC®), guided by the manipulator shaft as a landmark.
  Arms: laparoscopic isthmocele repair using Polyglactin 910 Vicryl sutures

SUMMARY:
To evaluate postoperative outcomes in patients with isthmocele undergoing laparoscopic repair, comparing the efficacy of V-LocTM 180 and Polyglactin 910 Vicryl sutures.

Patients were randomized to undergo laparoscopic isthmocele repair using one of the following suture materials: (1) V-LocTM 180 or (2) Polyglactin 910 Vicryl.

DETAILED DESCRIPTION:
The global rise in cesarean section (CS) rates has led to an increased incidence of associated complications, presenting new challenges in gynecological practice. One of these complications is a cesarean scar defect, also known as isthmocele, which manifests as a pouch-like structure at the site of the previous CS scar. This defect often results in the accumulation of menstrual blood, inflammatory cells, and mucus, leading to symptoms such as postmenstrual bleeding, pelvic pain, and dyspareunia. Furthermore, isthmocele has been implicated in secondary infertility due to the inflammatory changes it induces in the endometrium. Additionally, the presence of an isthmocele increases the risk of complications in future pregnancies, including cesarean scar ectopic pregnancy, uterine rupture, and placenta accreta spectrum disorders.

Diagnosis of isthmocele relies on imaging modalities such as transvaginal ultrasound (TVUS), sonohysterography (SHG), or hysteroscopy. While asymptomatic cases generally do not require intervention, symptomatic patients may benefit from medical or surgical treatment. Due to limited evidence supporting medical therapy, surgical intervention has become the preferred approach, particularly for patients desiring future fertility. Various surgical techniques, including hysteroscopic, laparoscopic, vaginal, laparotomic, and combined procedures, have been proposed for isthmocele repair. Among these, laparoscopic isthmocele repair is favored for patients with fertility concerns as it enables complete excision of the defective myometrial tissue and reconstruction of the uterine wall.

Despite the advantages of laparoscopic isthmocele repair, no universally accepted cutoff value for residual myometrial thickness dictates surgical candidacy. Previous studies have suggested that laparoscopic repair is a safer and more practical option for cases with significant myometrial loss (>80%). However, there is limited data on the impact of different suture materials used in laparoscopic repair on postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The study will include women aged 18-45 years who present with symptomatic isthmocele.
* Participants must have a residual myometrial thickness of less than 2.5 mm.
* Participants must desire future fertility.

Exclusion Criteria:

Age below 18 or above 45 years

Atypical endometrial cells or cervical dysplasia on cytology

Asymptomatic isthmocele

Candidacy for hysteroscopic surgery

Cervical or pelvic infections

Cervical dilation of 4 cm or more (emergency surgery)

Conditions impairing tissue healing, such as:

Type 1 or Type 2 diabetes mellitus

Hematologic disorders associated with bleeding diathesis

Contraindications for spinal or general anesthesia

Continuous use of oral contraceptives (OCPs) or GnRH agonists that affect menstrual cycles

Hydrosalpinx communicating with the uterine cavity

Intrauterine device (IUD) in place

Known connective tissue disorders

Menstrual irregularities:

Cycles longer than 35 days

Cycle variations of 2 weeks or more

Ongoing pregnancy

Presence of structural abnormalities such as:

Uterine or cervical polyps

Submucosal fibroids

Other similar conditions

Residual myometrial thickness > 2.5 mm

Retained placental tissue

Suspected malignancies

Uterine anomalies

Immunosuppressive diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Post-operative residual myometrial thickness | 1 year
  Ultrasonographic evaluation will be performed in the 12th postoperative month to measure residual myometrial thickness and assess the anatomical success of the repair.

SECONDARY OUTCOMES:
Patient satisfaction and quality of life | 1 year
  Participants will complete the Female Sexual Function Index (FSFI) questionnaire in the postoperative 12th month to evaluate sexual function and overall health-related quality of life.
3.Patient satisfaction | 1 year
  Participants will complete the SF-36 questionnaire in the postoperative 12th month to evaluate sexual function and overall health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No